CLINICAL TRIAL: NCT01863394
Title: Evaluation of Two Community Based Screening Strategies for Severe Acute Malnutrition in Children Aged 6-59 Months in the Mirria District, Niger
Brief Title: Evaluation of Two Community Based Screening Strategies for Severe Acute Malnutrition in Children 6-59 Months in Mirria District, Niger
Acronym: MàLÉ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for International Medical Action (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MUAC À L'ÉCHELLE
Record Dates: First submitted 2013-05-07; First posted 2013-05-29 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Malnutrition
Keywords: Screening; Malnutrition; Community Management of Acute Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Screening by community health workers (Active Comparator): One Community Health Worker (CHW) will be trained per village in the comparator arm. The training the CHWs receive will be identical to that delivered in the Community Management of Acute Malnutrition program run by ALIMA/BEFEN (Bien Être de la Femme et l'Enfant Niger) over the last 3 years. This involves 6 hours theoretical training and a practical session in the health centre.
  CHWs will screen children 06-59 months in their village once a month
  Interventions: Other: Active comparator: Screening by community health workers
- Screening by mothers (Experimental): Mothers in the intervention health district will be trained in small womens' groups in their village. Training will have a theoretical component and a practical demonstration component on children in the village
  During the first baseline door to door mass screening campaign, mothers will also receive individual training on conducting a Mid Upper Arm Circumference (MUAC) classification and looking for pedal oedema. they will receive a brief recap during the three monthly door-to-door mass screening campaigns
  Mothers will be asked to check their child's MUAC and look for pedal oedema
  * whenever the child does not seem to be in 'good health' to the mother
  * whenever the mother feels that the child is 'unwell' or 'sick'
  * whenever it seems to the mother that her child has lost weight
  * whenever the mother thinks that it is necessary to do so
  Interventions: Other: Screening by mothers

INTERVENTIONS:
Other: Screening by mothers
  Arms: Screening by mothers
Other: Active comparator: Screening by community health workers
  Arms: Screening by community health workers

SUMMARY:
The objective of this study is to determine the efficacity of a community strategy for screening children 06-59 months old for Severe Acute Malnutrition (SAM) conducted by their mothers' compared with a community screening strategy conducted by Community Health Workers.

ELIGIBILITY:
Inclusion Criteria:

* children aged 06-59 months at the time of the study
* children who live in a village in the health district participating in the study

Exclusion Criteria:

* children whose legal guardian refuses to participate in the study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4429 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The coverage of the therapeutic nutritional program in the control and intervention health districts | 12 months
  Coverage of the the therapeutic nutritional treatment program is defined as the proportion of children 06-59 months with Severe Acute Malnutrition (Mid Upper Arm Circumference <115mm and/or oedema) receiving treatment in the program, amongst the total number of children diagnosed with Severe Acute Malnutrition

SECONDARY OUTCOMES:
Malnutrition program data for children referred by community health workers & mothers | 12 months
  Nutritional status at admission (mid upper arm circumference +/- oedema) Type of admission to the programme (out-patient or immediate transfer for in-patient care) Source of reference to the programme (Community Health Worker, Mother, other) Date of discharge from the programme Weight at admission to the programme Discharge criteria (cured, died, failed to attend, non-response to treatment, transfer for in-patient nutrition care, transfer to other health care structures) Number of children screened by mothers confirmed to have SAM at the treatment centre Number of children screened by community health workers confirmed to have SAM at the treatment centre

CONTACTS AND LOCATIONS:
Overall Officials: Nikki BLACKWELL, FCICM, Principal Investigator — Alliance for International Medical Action; Isabelle Defourney, MBBS, Study Director — Alliance for International Medical Action
Locations (1):
- Mirriah health district, Mirriah, Zinder Region, Niger

REFERENCES:
- [Derived] Ale FG, Phelan KP, Issa H, Defourny I, Le Duc G, Harczi G, Issaley K, Sayadi S, Ousmane N, Yahaya I, Myatt M, Briend A, Allafort-Duverger T, Shepherd S, Blackwell N. Mothers screening for malnutrition by mid-upper arm circumference is non-inferior to community health workers: results from a large-scale pragmatic trial in rural Niger. Arch Public Health. 2016 Sep 6;74(1):38. doi: 10.1186/s13690-016-0149-5. eCollection 2016. PMID 27602207